CLINICAL TRIAL: NCT03666871
Title: T-Cell Reinfusion After Interfering With Lymphocyte Binding Location of AIDS Virus Through Zinc-finger-nuclease Elimination of CCR5 Receptors: The TRAILBLAZER Study
Brief Title: CCR5-modified CD4+ T Cells for HIV Infection
Acronym: TRAILBLAZER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: University of California, San Francisco (Other); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Carl J. Fichtenbaum, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRAILBLAZER
Record Dates: First submitted 2018-09-07; First posted 2018-09-12 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Arm 1 (n=20) will be pretreated with cyclophosphamide 1 g/m2 and will receive a single intravenous infusion of 0.5 to 4x1010 ex vivo expanded autologous CD4+ T cells that have been transduced with a zinc finger nuclease designed to cleave CCR5.
  Interventions: Biological: SB-728-T
- Arm 2 (Active Comparator): Arm 2 (n=10) will be pretreated with cyclophosphamide 1 g/m2 and will receive a single intravenous infusion of 0.5 to 4x1010 ex vivo expanded autologous CD4+ T cells that have not been modified by zinc finger nucleases.
  Interventions: Biological: Expanded unmodified autologous CD4+ T cells

INTERVENTIONS:
Biological: SB-728-T — Autologous CD4+ T cells with ex vivo modification of the CCR5 gene by zinc finger nucleases
  Arms: Arm 1
Biological: Expanded unmodified autologous CD4+ T cells — Autologous CD4+ T cells without ex vivo modification of the CCR5 gene by zinc finger nucleases
  Arms: Arm 2

SUMMARY:
A Comparative Study of Autologous CD4+ T Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases SB-728 versus ex vivo Expanded Unmodified Autologous CD4+ T Cells in Treated HIV-1 Infected Subjects

DETAILED DESCRIPTION:
This is a randomized clinical trial comparing the effect of infusing expanded autologous CD4+ T cells with or without ex vivo modification of the CCR5 gene by zinc finger nucleases among HIV-infected patients with plasma HIV RNA levels <50 copies/mL for at least 48 weeks and CD4+ T cell counts greater than 350 cells/µL. The main hypothesis is that the infusion of modified CD4+ T cells will lead to a reduction in the size of the replication-competent HIV reservoir, that is greater than that resulting from infusion of unmodified CD4+ T cells. A total of 30 participants will be randomized to receive one infusion of 0.5 - 4 x 1010 ex vivo expanded autologous CD4+ T cells that have been either modified by transduction with a zinc finger nuclease designed to cleave CCR5 (arm 1, n=20) or unmodified (arm 2, n=10). All participants will be pre-treated with cyclophosphamide at a dose of 1 g/m2 before infusion. The primary outcome measure the difference in the magnitude of change in intact provirus from before infusion to 96 weeks after infusion between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by study subject.
2. Men or women, including trans men or women, ≥18 and ≤70 years of age.
3. For persons born male who have not been surgically sterilized, willingness to abstain from sexual activity that could result in conception for 90 days after the cyclophosphamide administration visit.
4. HIV-1 infection, documented by any FDA-approved ELISA, EIA, or rapid antibody detection method, and confirmed by a second FDA-approved antibody-based test or by a positive FDA-approved HIV RNA detection assay. FDA-approved HIV-1 RNA detection assay alone constitutes proof of HIV-1 infection assuming there is documentation of >199 copies/mL of HIV-1 RNA in the absence of antiretroviral therapy.
5. Adequate venous access for leukapheresis, as documented by standard clinical procedures at each site.
6. The following laboratory values at screening:

   1. Absolute neutrophil count (ANC) > 1500/mm3
   2. Hemoglobin level ≥11 g/dL
   3. Platelet count ≥150,000/mm3
   4. Serum creatinine <1.5 mg/dL
   5. AST and ALT ≤2.5 times the upper limit of normal
   6. CD4+ T cell count > 350 cells/mm3
   7. HIV-1 RNA <50 copies/mL performed with an ultrasensitive HIV-1 PCR assay.
   8. Urine red blood cell (RBC) counts within the normal range used by each institution.
   9. INR ≤1.5 and PTT ≤2xULN
7. Willing to comply with study-mandated evaluations.
8. All participants must have received combination antiretroviral therapy, and had plasma HIV RNA levels <50 copies/mL for at least 48 weeks. Subjects who had intermittent isolated episodes of detectable low-level viremia <500 copies RNA/mL flanked by values <50 copies/mL will remain eligible.
9. On stable antiretroviral medication (no changes to treatment and no missed dose for >7 continuous days within 4 weeks of screening) and willing to continue on current antiretroviral therapy, unless a change is medically indicated, for the duration of the study. Note: Changes in formulation or a single within-class, single-agent change are permitted in the last 48 weeks but not within 12 weeks of study entry.

Exclusion Criteria:

1. Women and persons born female regardless of gender identity with childbearing potential. These participants are considered to be of childbearing potential if they are postmenarchial, have an intact uterus and at least one ovary, and have had at least one menstrual period in the past two years. Participants who have had a documented bilateral tubal ligation or a hysterectomy are not considered to be of childbearing potential.
2. Previous gene therapy using an integrating vector. NOTE: For the purposes of the TRAILBLAZER protocol, only therapies that a) are expected to modify the host genome durably or broadly, and b) are delivered using a vector defined by FDA as having a propensity for integration or the potential for latency/reactivation meet this exclusion criterion. The following are examples of products and vectors that DO NOT meet this exclusion criteria:

   * Plasmid DNA products
   * RNA products
   * Poxvirus-vectored products
   * Adenovirus-vectored products
   * Replication-negative adeno-associated virus-vectored products
   * Prophylactic or therapeutic HIV vaccines that use one of these delivery mechanisms
3. Allergy or hypersensitivity to study product excipients (human serum albumin, DMSO and Dextran 40).
4. An antiretroviral regimen including maraviroc or any CCR5 inhibitor within 4 weeks prior to screening.

   Presence or absence of the following exclusion criteria will be assessed at screening, but participants who develop any of these criteria at any time between screening and the planned infusion time will be excluded:
5. Acute or chronic hepatitis C infection, defined as a positive plasma HCV RNA using any FDA-approved qualitative or quantitative test in a participant with a positive HCV antibody (HCV RNA testing is not required in participants with a negative HCV antibody) at screening. Participants who have completed a course of antiviral treatment for hepatitis C and have a confirmed plasma HCV RNA level below the limit of detection of the assay 12 weeks or longer after completion of therapy will be eligible. Note: Individuals that have undetectable HCV RNA in the absence of treatment that cleared infection spontaneously are also considered eligible to participate.
6. Acute or chronic hepatitis B infection, defined as a positive HBV surface antigen or a positive HBV DNA at screening.
7. Any prior AIDS-defining condition within the past 5 years, except a history of CD4+ T cell count below 200 cells/mm3.

   NOTE: The terms "AIDS encephalopathy" and "wasting syndrome" are often recorded on medical records to indicate constellations of signs and symptoms that may not formally meet the current diagnostic criteria for AIDS-related dementia or AIDS-associated wasting syndrome, respectively. Therefore, the principal investigators will determine whether in their opinion, a reported history of these conditions truly corresponds to an AIDS-defining syndrome meeting this criterion.
8. Any active cancer or malignancy within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin or low-grade (0 or 1) anal or cervical intraepithelial neoplasia.
9. Diagnosis of New York Heart Association (NYHA) grade 3 or 4 congestive heart failure, uncontrolled angina or uncontrolled arrhythmias.
10. Corrected QT interval (QTc) >470 msec (by any formula).
11. History or any features on physical examination indicative of a bleeding diathesis.
12. Use of chronic corticosteroids, hydroxyurea, or immune-modulating agents (e.g., interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to screening or for any period extending to within 30 days prior to the planned infusion date.

    NOTE: Use of inhaled or topical steroids is not exclusionary.
13. Breastfeeding or pregnant.
14. Continued need for use of aspirin, warfarin or any other medication likely to affect platelet function or other aspects of blood coagulation significantly that cannot be held during the 7-day period prior to each of the leukapheresis procedures (or tissue/CSF sampling procedures for participating subjects) or that maintains biological activity beyond 7 days after discontinuation.
15. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
16. Presence at screening of a serious and persistent illness requiring a new systemic treatment expected to last beyond the planned date of infusion and/or hospitalization within 30 days prior to the planned date of infusion.

    NOTE: A participant who has required a hospital admission within the 30 days prior to infusion may be allowed to proceed if, in the judgement of the principal investigators, the condition requiring admission has resolved completely and is not expected to recur or worsen during study participation. Examples include scenarios such as: a removed kidney stone; inpatient hydration for food poisoning; observation for atypical chest pain; a minor traumatic injury; etc.
17. Planned or actual vaccine administration within 4 weeks prior to infusion. Note: Receipt of a COVID-19 vaccine authorized under an FDA EUA, in general, should not disqualify potential participants. Vaccination should be avoided in the 4 weeks prior to and after the administration of cyclophosphamide. In addition, vaccination should be avoided 2 weeks prior to study leukapheresis or large volume blood draw.
18. Intercurrent illness that in the opinion of the investigator may compromise the safety of the participant or interfere with study objectives.
19. Current use of zidovudine within 30 days of planned infusion of cyclophosphamide.
20. Current active chronic liver disease (e.g., cirrhosis or non-alcoholic steatohepatitis) within 30 days of study enrollment. Note: In addition, for the purpose of the TRAILBLAZER clinical trial, chronic active liver disease means a confirmed diagnosis of cirrhosis of the liver or non-alcoholic steatohepatitis with elevated liver transaminases (confirmed) above the upper limit of normal. The presence of fat (steatosis or NAFLD) in the liver by imaging (in the absence of indication of disease, e.g., elevated transaminases) is not a contraindication to enrollment in the trial. Individuals diagnosed with fatty liver disease that have normal transaminases may be permitted to enroll in the study. The use of FDA approved medications to treat chronic fatty liver disease is a contraindication to enrollment. The use of non-FDA approved interventions, vitamins or supplements is not a contraindication to enrollment.
21. A history of urinary outflow obstruction as documented by a history of enlarged prostate on physical exam, use of medications to treat outflow obstruction (e.g., tamsulosin), or elevated urinary residual volume. Note: urinary outflow obstruction is defined as requiring placement of a drainage catheter to relieve a urinary obstruction. Documented enlargement of the prostate in the absence of urinary obstruction is not a contraindication to enrollment in the trial. The use of FDA approved medications to treat urinary frequency (e.g., tamsulosin) in the absence of proven urinary obstruction is not a contraindication to enrollment.
22. A history of active or latent tuberculosis, regardless of treatment history.
23. Individuals with limited antiretroviral treatment options (less than 2 new classes) by history because of prior known resistance mutations to antiretrovirals. Note: Investigators should consider prior treatment history for HIV and known resistance mutations to ensure that a potential participant has an acceptable alternative treatment regimen should they develop treatment failure while on study.
24. Inability, in the opinion of the investigator, to avoid potential exposure to Covid-19 in the two weeks after the receipt of cyclophosphamide. Note: Participants may go out into public to conduct essential activities but will be strongly encouraged to wear a mask, use appropriate social distancing and hand hygiene when going outside their home during that 14 day interval.
25. Any other condition that, in the opinion of the clinical investigator or sponsor, might compromise any aspect of this trial.

For participants in the rectosigmoid biopsy program only:

1. Major GI tract surgery within 45 days prior to the planned date of the baseline visit. Minor procedures involving only the anal canal such as condyloma ablations, hemorrhoidectomy, and anoscopy are permitted if cleared by the responsible surgeon.
2. Abnormalities of the colorectal mucosa, or significant colorectal symptoms, which in the opinion of the clinician represent a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa).

For participants in the lymph node biopsy program at sites doing open biopsies only:

1. BMI greater than 35 at screening.
2. Anatomical condition that would prevent surgical access to either inguinal area, such as scar tissue, active skin condition affecting the area, or foreign material.
3. Known hypersensitivity to local anesthetic agents.
4. Contraindication for the use of epinephrine-containing local anesthetic formulations.
5. Presence of pacemaker, implantable defibrillator, or other medical device thought to be susceptible to electromagnetic interference from electrocautery.

For participants in the lymph node biopsy program at sites doing lymph node aspirates only:

1. Anatomical condition that would prevent surgical access to either inguinal area, such as scar tissue, active skin condition affecting the area, or foreign material.
2. Known hypersensitivity to local anesthetic agents.
3. Contraindication for the use of epinephrine-containing local anesthetic formulations.

For participants in the CSF sampling program only:

1. Any condition that could prevent access to the subarachnoid space or obscure the anatomical landmarks for lumbar puncture, such as scar tissue, active skin condition affecting the area, or foreign material.
2. Known hypersensitivity to local anesthetic agents.
3. Known space-occupying central nervous system lesion, unless cleared by the treating physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Difference in the magnitude of change in intact provirus from before infusion to 96 weeks after infusion between the two study arms. | 96 weeks
  Difference in the magnitude of change in intact provirus from before infusion to 96 weeks after infusion between the two study arms.
Difference in the proportion of participants who experience a grade ≥3 adverse event that is considered possibly, probably, or definitely related to study treatment between the two study arms. | 96 weeks
  Difference in the proportion of participants who experience a grade ≥3 adverse event that is considered possibly, probably, or definitely related to study treatment between the two study arms.
Proportion of participants who experience a grade ≥3 adverse event that is considered possibly, probably, or definitely related to study treatment in each of the study arms. | 24 months
  Proportion of participants who experience a grade ≥3 adverse event that is considered possibly, probably, or definitely related to study treatment in each of the study arms.

SECONDARY OUTCOMES:
Difference in the magnitude of change in intact provirus from before infusion to 48 weeks after infusion between the two study arms. | 48 weeks
  Difference in the magnitude of change in intact provirus from before infusion to 48 weeks after infusion between the two study arms.
Change in the log10 copy-number of intact proviruses per million CD4+ T cells from the first leukapheresis visit to the week 48 visit. | 48 weeks
  Change in the log10 copy-number of intact proviruses per million CD4+ T cells from the first leukapheresis visit to the week 48 visit.
Change in the log10 copy-number of intact proviruses per million CD4+ T cells from the first leukapheresis visit to the week 96 visit. | 96 weeks
  Change in the log10 copy-number of intact proviruses per million CD4+ T cells from the first leukapheresis visit to the week 96 visit.
Peripheral CD4+ T cell count at each of the follow-up time points after infusion of ex vivo expanded CD4+ T cells in each study arm. | 96 weeks
  Peripheral CD4+ T cell count at each of the follow-up time points after infusion of ex vivo expanded CD4+ T cells in each study arm.
Frequency of pentamer PCR-positive CD4+ T cells in peripheral blood at each of the follow-up time points after infusion of ex vivo expanded CD4+ T cells in the CCR5-modified study arm | 96 weeks
  Frequency of pentamer PCR-positive CD4+ T cells in peripheral blood at each of the follow-up time points after infusion of ex vivo expanded CD4+ T cells in the CCR5-modified study arm
Frequency of pentamer PCR-positive CD4+ T cells in cell suspensions of rectal biopsy tissue | 96 weeks
  Frequency of pentamer PCR-positive CD4+ T cells in cell suspensions of rectal biopsy tissue
Frequency of pentamer PCR-positive CD4+ T cells in cell suspensions of lymph node biopsy tissue | 96 weeks
  Frequency of pentamer PCR-positive CD4+ T cells in cell suspensions of lymph node biopsy tissue
Frequency of pentamer PCR-positive CD4+ T cells in CSF | 96 weeks
  Frequency of pentamer PCR-positive CD4+ T cells in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Carl Fichtenbaum, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared once primary and secondary manuscripts are completed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After acceptance of primary and secondary manuscripts. Available for 3 years after above.
Access Criteria: Contact the Study Principal investigator to obtain information. Requests will be reviewed by the core team for approval.